CLINICAL TRIAL: NCT06755996
Title: Combination of Dexmedetomidine Nasal Spray and Remimazolam for the Treatment of Pediatric Bronchoscopy
Brief Title: Dexmedetomidine Nasal Spray and Pediatric Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEXS
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Fiberoptic Bronchoscopy
MeSH Terms: interventions — Dexmedetomidine; remimazolam

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DR1 group (Active Comparator): Dexmedetomidine injection 3μg/kg+ remimazolam 0.5mg/kg group
  Interventions: Drug: Dexmedetomidine injection; Drug: Remimazolam
- DR2 group (Experimental): Dexmedetomidine nasal spray 3μg/kg+ remimazolam 0.5mg/kg group
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Dexmedetomidine injection — Dexmedetomidine injection 3μg/kg
  Other Names: dex inj
  Arms: DR1 group
Drug: Remimazolam — remimazolam 0.5mg / kg
  Other Names: remi

SUMMARY:
To observe the sedative effect of using dexmedetomidine nasal spray combined with remimazolam for pediatric bronchoscopy diagnosis and treatment, provide a safer and more comfortable anesthesia plan for pediatric bronchoscopy diagnosis and treatment

DETAILED DESCRIPTION:
Dexmedetorimidine nasal spray is a new dosage form, which is simple and easy to achieve sedative and anti-anxiety effects by nasal spray mucosa. In the dose range from 50 to 100 μ g, the sedation effect increased dose-dependent, with> 2 μ g / kg administered, and the child could be successfully separated within 45min.Our study is to observe the sedative effect of using dexmedetomidine nasal spray combined with remimazolam for pediatric bronchoscopy diagnosis and treatment, provide a safer and more comfortable anesthesia plan for pediatric bronchoscopy diagnosis and treatment

ELIGIBILITY:
Inclusion Criteria:

* Age 2-6 years old (24~72 months);
* ASA I-II;
* sign the informed consent.

Exclusion Criteria:

* Severe rhinitis, nasal deformity;
* abnormal liver and kidney function;
* severe dehydration, severe malnutrition, hypoproteinemia or anaemia Hb <10 g/dl;
* children with neurological disease;
* history of allergy to the study drug;
* recent participation in other clinical studies.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Sedation success rate | 1day
  MOSS / A score =4-point time

SECONDARY OUTCOMES:
recoving time | 1day
  Wake up time
Drug dosage | 1day
  dosage of dexmeditomidine and remimazolam

CONTACTS AND LOCATIONS:
Overall Officials: pu zhou, Dr., Study Chair — Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No